CLINICAL TRIAL: NCT05465590
Title: A Phase 1 Study to Evaluate the Pharmacokinetics and Safety of MB1707 in Patients With Advanced Cancer
Brief Title: A Phase 1 Study to Evaluate Paclitaxel Conjugated CXC Receptor 4 Antagonist (MB1707) in Patients With Advanced Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to Sponsor decision
Sponsor: Mainline Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLB-PK-001
Record Dates: First submitted 2022-07-16; First posted 2022-07-20 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor; Breast Cancer; Non Small Cell Lung Cancer; Ovary Cancer; Pancreatic Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MB1707 Single Dose Phase 1 (Experimental): Phase 1 MB1707 given as a single intravenous (IV) dose of 0.3 mg/kg
  Interventions: Drug: MB1707

INTERVENTIONS:
Drug: MB1707 — MB1707 is a CXCR4 antagonist peptide-conjugated paclitaxel.
  MB1707, paclitaxel (PTX) conjugated CXC chemokine receptor 4 (CXCR4) peptide antagonist, a peptide-drug conjugate (PDC), for the treatment of cancer. MB1707 is a potent CXCR4 antagonist which inhibits tumor growth and metastasis by blocking the stromal cell derived factor 1 (SDF-1, a.k.a. CXCL12)/CXCR4 signaling pathway. MB1707 contains a conjugated drug, paclitaxel. By specific binding to CXCR4 overexpressed by the tumor cells, MB1707 has a built-in targeted delivery mechanism.

SUMMARY:
The study will evaluate the pharmacokinetics (PK) and safety of a single intravenous (IV) dose of 0.3 mg/kg MB1707 in patients with advanced cancers.

DETAILED DESCRIPTION:
MB1707, paclitaxel (PTX) conjugated CXC chemokine receptor 4 (CXCR4) peptide antagonist, a peptide-drug conjugate (PDC), for the treatment of cancer. MB1707 is a potent CXCR4 antagonist which inhibits tumor growth and metastasis by blocking the stromal cell derived factor 1 (SDF-1, a.k.a. CXCL12)/CXCR4 signaling pathway. MB1707 contains a conjugated drug, paclitaxel. By specific binding to CXCR4 overexpressed by the tumor cells, MB1707 has a built-in targeted delivery mechanism.

The study will evaluate the PK and safety of a single intravenous (IV) dose of 0.3 mg/kg MB1707 in patients with advanced cancers.

Up to 6 patients will be enrolled.

Patients will be treated with a single intravenous (IV) dose of MB1707 over 3 hours on Day 1 only.

Patients will be pre-medicated with an antihistamine (eg, diphenhydramine), a corticosteroid (e.g., dexamethasone), and a H2 receptor antagonist (e.g., famotidine), within 30 to 60 minutes prior to infusion at doses per institutional guidelines.

Patients will be observed for 60 minutes after Cycle 1 dose administration.

Patients will complete a 14-day Safety Follow-up Visit following the single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥18 years at the time of informed consent.
2. Patients who have previously received at least one line of standard systemic therapy for their advanced/metastatic cancer and have either progressed, recurred, or were intolerant to the previous treatment eligible for treatment with a paclitaxel-based regimen.
3. Clinical Performance Status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
4. Adequate bone marrow reserves
5. Adequate major organ system function
6. Female patients must not be pregnant or breastfeeding.

Exclusion Criteria:

1. Patients with tumor primarily localized to the brainstem or spinal cord. Presence of known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth.
2. Patients with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
3. Patients with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
4. Major surgery within 4 weeks prior to study entry.
5. Systemic anticancer therapy within 4 weeks prior to study entry
6. Bleeding esophageal or gastric varices <2 months prior to the date of informed consent.
7. History of severe immediate hypersensitivity reaction to paclitaxel
8. Active unstable or clinically significant medical condition
9. History of any major cardiovascular conditions within the past 6 months
10. Patients with known active, uncontrolled bacterial, fungal, or viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) as characterized by type, frequency, severity (NCI CTCAE Version 5.0), timing, seriousness, and relationship to study therapy | 14 days
  Treatment-emergent AEs through 14 days after last protocol therapy will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) Version 14.0 (or higher) System Organ Class and preferred term. The incidences and percentages of participants experiencing each AE preferred term will be summarized with descriptive statistics. AEs will also be summarized by NCI CTCAE, Version 5.0, by grade and by causality (attribution to study treatment).
Peak Plasma Concentration (Cmax) | 2 days
  Determine Maximum observed MB1707 concentration from the time of dosing (0 h) to the time of the last quantifiable MB1707 concentration following dose administration
Time to Cmax (Tmax) | 2 days
  Determine Time of maximum observed MB1707 concentrations (post-dose)
Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) | 2 days
  Determine Area under the MB1707 concentration-time curve from the time of dosing (0 h) to the time of the last quantifiable concentration following dose administration
Area under the concentration-time curve extrapolated to infinity (AUC∞) | 2 days
  Determine Area under the MB1707 concentration-time curve from the time of dosing (0 h), extrapolated to infinity
Half-life in plasma (t1/2) | 2 days
  Determine Apparent terminal phase half-life of MB1707
Total body clearance (CL) | 2 days
  Determine total body clearance MB1707
Volume of distribution (VZ) | 2 days
  Determine Volume of distribution based on the terminal Phase of MB1707

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Weitzman, MD, Study Director — Mainline Biosciences

IPD SHARING:
Plan to Share IPD: No